CLINICAL TRIAL: NCT03442907
Title: Intraoperative Blood Pressure Management Based on the Individual Blood Pressure Profile: Impact on Postoperative Organ Function
Brief Title: Personalized Blood Pressure Management
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMPROVE-1.0
Record Dates: First submitted 2018-01-19; First posted 2018-02-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Blood Pressure; Intraoperative Hypotension; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Fluid Therapy; Vasoconstrictor Agents; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The intraoperative blood pressure target for all patients in the study group is the mean arterial pressure (+ 10mmHg maximum) derived from the prior 24-hour blood pressure measurement.
  To achieve the blood pressure target, fluid or vasoactive substances will be used.
  Interventions: Procedure: 24 hour blood pressure measurement, fluids, vasopressors
- Control group (Active Comparator): Study patients of the control group are treated according to the standard operating procedures (SOP) of the Department of Anaesthesiology, University Medical Centre Hamburg Eppendorf.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: 24 hour blood pressure measurement, fluids, vasopressors — Targeting individual blood blood pressure values during surgical procedures
  Arms: Study group
Procedure: Standard of Care — Treatment according to Standard of care at the Department of Anaesthesiology, University Medical Centre Hamburg Eppendorf
  Arms: Control group

SUMMARY:
The aim of this research project is to find out whether a personalized definition of the lower blood pressure threshold based on the individual blood pressure profile by means of preoperative 24-hour blood pressure measurement can reduce organ damage (brain, kidney, heart) through reduced blood flow during surgery.

ELIGIBILITY:
Inclusion Criteria

* age ≥ 50 years
* ASA II-IV (Classification of the American Society of Anesthesiologists for the assessment of the perioperative risk depending on the underlying diseases)
* duration of intervention in general anesthesia at least 90 minutes

Exclusion Criteria:

* Pregnancy
* Emergency procedures
* Surgery requiring controlled hypotension (e.g., aneurysm)
* Cerebrovascular events in the past medical history
* Patients of cardiac surgery, vascular surgery, neurosurgery, and transplantation surgery
* Pre-existing dementia (anamnesis)
* kidney transplant
* dialysis-dependent renal insufficiency (KDIGO criteria)
* no patient consent
* failure to meet the inclusion criteria
* Impossibility of 24-h blood pressure measurement

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Composite endpoint: Incidence of POCD or delirium | 3rd-7th postoperative day
  POCD is measured on the basis of a neuropsychological test battery and the delirium on the basis of the CAM-ICU test.

SECONDARY OUTCOMES:
Kidney function | 24, 48 and 72 hrs after surgery
  Glomerular filtration rate; calculated 24h, 48h and 72h after surgery (Cockcroft-Gault equation)
cardiac ischemia | 6 hours after surgery
  high-sensitive troponin T measurements are performed prior and 6 hours after surgery
length of hospital stay | 30 days
30-day mortality | 30 days
30-day morbidity | 30 days
  European perioperative outcome definitions

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Anästhesiologie, Zentrum für Anästhesiologie und Intensivmedizin, Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Nicklas JY, Bergholz A, Dake F, Pham HHD, Rabe MC, Schlichting H, Skrovanek S, Flick M, Kouz K, Fischer M, Olotu C, Izbicki JR, Mann O, Fisch M, Schmalfeldt B, Frosch KH, Renne T, Krause L, Zollner C, Saugel B. Personalised blood pressure management during major noncardiac surgery and postoperative neurocognitive disorders: a randomised trial. BJA Open. 2024 Jul 1;11:100294. doi: 10.1016/j.bjao.2024.100294. eCollection 2024 Sep. PMID 39050403